CLINICAL TRIAL: NCT05578534
Title: CO2 Gap Changes Compared to Cardiac Output Changes in Response to Intravenous Volume Expansion and/or Vasopressor Therapy in Septic Shock
Brief Title: CO2 Gap Changes in Septic Shock in Relation to Cardiac Output
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mostafa Farouk, Lecturer of critical care, Cairo University
Other Study IDs: MD-194-2019
Record Dates: First submitted 2022-10-05; First posted 2022-10-13 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Septic Shock
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 28 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- High CO2 gap (Pcv-aCO2 > 6 mmHg): Patients had high PCO2 gaps before initial resuscitation
- Normal CO2 gap (Pcv-aCO2 ≤6 mmHg): Patients had normal PCO2 gaps before initial resuscitation
- Responsive (15% increase in CI or stable MAP was achieved): Patients who respond to initial resuscitation with 15% increase in CI
- Non-responsive (< 15% increase in CI or a stable MAP was not achieved): Patients who do not respond to initial resuscitation with less than 15% increase in CI
- Survivors: Patients who survived after 28 days
- Non survivors: Patients who do not survive within 28 days

SUMMARY:
Background The arteriovenous difference of partial pressure of carbon dioxide (PCO2) between mixed or central venous blood and arterial blood is the ∆PCO2 or CO2 gap. Previous data demonstrated a strong relationship between ∆PCO2 and cardiac index (CI) at the very early phase of resuscitation in septic shock. Monitoring the ∆PCO2 from the beginning of the resuscitation may be a useful tool to assess the adequacy of cardiac output (CO) in tissue perfusion.

Aim of work: To examine behavior of ∆PCO2 during early management of septic shock.

Methodology: Seventy-six patients with diagnosis of septic shock admitted to critical care department, Cairo university hospitals. We classified the study population according to initial resuscitation response, initial CO2 gap, or 28-days mortality. The response vs non-response to initial resuscitation, ICU morbidity and recovery rate were the study primary outcomes while secondary outcomes included ICU length of stay (LOS) and 28-day ICU Mortality.

DETAILED DESCRIPTION:
Introduction

Shock is defined as a life-threatening, generalized acute circulatory failure with inadequate cellular oxygen utilization [1]. One of the goals of acute circulatory failure treatment is to increase cardiac output [2].

The ∆PCO2 is defined by the difference in the partial pressure of carbon dioxide (PCO2) between mixed or central venous blood and arterial blood [1]. The ∆PCO2 has been correlated to outcome and mortality [3].

The mixed ∆PCO2 difference has been shown to be inversely correlated with the cardiac index (CI). A central venous PCO2, which is easier to obtain, may provide similar information. Substitution of a central for a mixed ∆PCO2 provides an accepted alternative [4].

Measurements of central venous oxygen saturation (ScvO2) and ∆PCO2 were advised to assess adequacy of cardiac output as well as to guide therapy [5]. A normal CO2 gap indicates that CO is high enough to wash out CO2 from peripheral tissue. Either PCO2 gap or the PCO2 gap to arterio-venous O2 content difference ratio could be used to guide resuscitation therapy [6].

∆PCO2 value of >6 mmHg suggests an insufficient blood flow in the tissues even when the ScvO2 is >70 % [1].

Aim of work

Our aim of the study is to investigate the value of PCO2 gap changes in the early septic shock management compared to the cardiac output.

Patients and methods

The study was approved by the ethical committee of faculty of medicine, Cairo University (N-194-2019)

A written informed consent was obtained from patient's first degree relatives.

Sample size calculation Based on past review of literature and by using G power software (version 3.1.3, Heinrich-Heine-Universität, Düsseldorf Germany) with a power of 0.90 and 0.05 alpha error, sample size was calculated to be 69 patients. With a withdrawal/non-evaluable subject rate of 10%, a total of 76 patients will be recruited.

Type of the study An observational prospective study was conducted on 76 consecutive adult patients admitted to critical care department of Cairo university hospitals with septic shock and elevated blood lactate level > 2 mmol/ L requiring fluid resuscitation and/ or vasopressor drugs infusion.

Duration : between December 2020 to March 2022

Definitions

Sepsis is identified by suspected or confirmed infection AND an organ dysfunction as defined by a sequential organ failure assessment (SOFA) [7].

Organ dysfunction defined by an increase in SOFA score of 2 points or more (sepsis-related) from up to 48 hours before to up to 24 hours after the onset of suspected infection [8].

Septic shock is clinically identified by a vasopressor requirement to maintain a mean arterial pressure of 65 mm Hg or greater and serum lactate level greater than 2 mmol/L (>18 mg/dL) in the absence of hypovolemia [7].

Inclusion criteria The study population were included immediately on admission to ICU after fulfilling inclusion criteria.

Exclusion criteria Patients with advanced cardiac, pulmonary, hepatic, or renal diseases were excluded from enrolment.

Our patients were resuscitated according to surviving sepsis campaign recommendations within 1 hr of recognition. The study cohort were included immediately on admission to ICU and after insertion of invasive lines (T0).

The resuscitation targets were MAP ≥ 65 mmHg, urine output ≥ 0.5 ml/kg/min, ScvO2 ≥ 70%, normalization or significant decrease of serum lactate concentration.

Infusion of vasopressors during or after fluid resuscitation if MAP cannot be maintained, and infusion of dobutamine if evidence of myocardial dysfunction or ongoing hypoperfusion despite optimizing intravascular volume.

The 1st set of measurements were taken after insertion of invasive lines (T0) & 2nd set of measurements were taken (T1) after completion the initial resuscitation when stable MAP by a fluid boluses of up to 30 ml/kg iv and/or by vasopressor infusion or after 3 hours which is closer.

Patients' demographics, comorbidities, APACHE II score up on ICU admission, SOFA score (initial and after 48 hrs), arterial lactate, ∆PCO2, blood gases (ABG, cvVBG), vital signs, echocardiographic LVOT cardiac output and index data were collected.

The microbiological data, source of sepsis, relevant laboratory data, vasopressor/inotropic support, ventilatory support, continuous renal replacement therapy (CRRT) needs along with ICU-morbidities and readmissions were recorded.

Lactate clearance was calculated as a percentage ratio of (initial arterial lactate level at T0 - arterial lactate level at 6 hours after treatment)/ arterial lactate level at T0. The P/F ratio, ∆PCO2 (before and after resuscitation), PCO2 Gap at T1/PCO2 Gap at T0 (gap/gap ratio) and cardiac index responsiveness was calculated as well.

The patients were classified according to initial ∆PCO2, resuscitation response, and 28-days mortality into:

1. High gap (Pcv-aCO2 > 6 mmHg) vs normal gap (Pcv-aCO2 ≤6 mmHg) [9] [10],
2. Responsive (15% increase in CI or stable MAP was achieved) vs non-responsive (< 15% increase in CI or a stable MAP was not achieved) [11] [12]
3. Survivors vs non-survivors

The gap/gap ratio is an expression of the trend of ∆PCO2 level during resuscitation and thus, it can be reflection of prognosis and outcome.

Response to resuscitation:

investigators defined the positive response to initial resuscitation as an increase in CI by 15% or a stable MAP was achieved within or after completion of the 1st 3 hrs post-enrolment. This cut-off value was chosen by the reference to previous studies.

ELIGIBILITY:
Inclusion Criteria:

* adult patients admitted to critical care department of Cairo university hospitals with septic shock and elevated blood lactate level > 2 mmol/ L requiring fluid resuscitation and/ or vasopressor drugs infusion.

Exclusion Criteria:

* Patients with advanced cardiac, pulmonary, hepatic, or renal diseases were excluded from enrolment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 76 consecutive adult patients admitted to critical care department of Cairo university hospitals with septic shock
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
The response to initial resuscitation | 6 hours
  response to intial resuscitation with IV fluids and vasopressors measured by PCO2 gap

SECONDARY OUTCOMES:
ICU length of stay (LOS) and 28-day mortality | 28 days
  correlation of measuring PCO2 gap as a resuscitation measure with ICU stay and mortality

CONTACTS AND LOCATIONS:
Overall Officials: Farouk Faris, MD, Principal Investigator — Cairo University
Locations (1):
- Critical care department, Cairo, Egypt